CLINICAL TRIAL: NCT05684263
Title: An Experimental Study of the Effects of Weight Science and Nutrition Education on Weight Control Beliefs and Disordered Eating in a Non-clinical Female Sample.
Brief Title: The Effects of Weight Science and Nutrition Education on Weight Control Beliefs and Disordered Eating.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Michele Laliberte, Psychologist, Clinical Lead, Eating Disorder Clinic, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STJOES2022WCB
Record Dates: First submitted 2022-11-29; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Body Image; Eating, Healthy
Keywords: Body Image; Weight control beliefs; Diet, Weight Loss; Eating, Healthy
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: There are three conditions in the study, which correspond to what education the participant will receive. The participant will be randomly assigned to one of the three conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Weight Science + Healthy Eating Education (Experimental): In this condition participants will watch two educational videos on the topics of weight science, and healthy eating. The videos were created by a registered psychologist and are each between 20 and 30 minutes in length.
  Interventions: Other: Weight Science Educational Video; Other: Healthy Eating Educational Video
- Weight Science + Healthy Sleep Education (Other): In this condition participants will watch two educational videos on the topics of weight science, and healthy sleep. The videos were created by a registered psychologist and are each between 20 and 30 minutes in length.
  We are interested in the effect of weight science education alone, the healthy sleep video was added as an active control so that each condition was watching the same amount of videos.
  Interventions: Other: Weight Science Educational Video; Other: Healthy Sleep Educational Video
- Healthy Eating + Healthy Sleep Education (Other): In this condition participants will watch two educational videos on the topics of healthy eating, and healthy sleep. The videos were created by a registered psychologist and are each between 20 and 30 minutes in length.
  We are interested in the effect of healthy eating education alone, the healthy sleep video was added as an active control so that each condition was watching the same amount of videos.
  Interventions: Other: Healthy Eating Educational Video; Other: Healthy Sleep Educational Video

INTERVENTIONS:
Other: Weight Science Educational Video — Educational videos on the topic of weight science created by a registered clinical psychologist.
  Arms: Weight Science + Healthy Eating Education; Weight Science + Healthy Sleep Education
Other: Healthy Eating Educational Video — Educational videos on the topic of healthy eating created by a registered clinical psychologist.
  Arms: Healthy Eating + Healthy Sleep Education; Weight Science + Healthy Eating Education
Other: Healthy Sleep Educational Video — Educational videos on the topic of healthy sleep created by a registered clinical psychologist.
  Arms: Healthy Eating + Healthy Sleep Education; Weight Science + Healthy Sleep Education

SUMMARY:
People have different beliefs about controlling their weight. Individuals who believe they should control their weight are more likely to have poor body image, low self-esteem and disordered eating. Individuals who believe they should aim for a healthy lifestyle and accept their natural weight have better body image, better self-esteem and less disordered eating. This study investigates the impact of three types of education on participants' beliefs about controlling weight: 1) education about the body's natural regulation of weight; or 2) education about healthy nutrition; or 3) education about both the body's regulation of weight and healthy nutrition. The study will also investigate whether changing participants' beliefs about controlling weight impacts participants' body satisfaction, feelings about themselves and intention to diet. It is predicted that teaching both about the body's regulation of weight and healthy eating will decrease participants' belief in personal control over weight, and increase participants' belief in striving for a healthy lifestyle and accepting their natural weight. In turn, these changes in weight control beliefs are expect to predict improved body satisfaction, feelings about themselves and a lower intention to diet.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of three conditions: 1) weight science + control (sleep education); 2) control (sleep education) + healthy nutrition education; or 3) weight science + healthy nutrition education. Participants will be randomly assigned to one of the three conditions by an algorithm in REDCap. The same procedure will be used for each condition, with the exception of what education is provided.

After the online consent form is completed, participants will be automatically redirected to the study questionnaires in REDCap. Participants will complete a package of questionnaires pre- and post- intervention measuring demographic information, physical activity, knowledge of weight science, weight control beliefs, self-esteem, restrained eating, body appreciation, self-compassion for weight and shape and fear of self-compassion for weight and shape. Participants will complete the package of questionnaires prior to watching two educational videos embedded into the REDCap project, and then complete the same package of questionnaires again.

After watching the educational videos and completing the study questionnaires, participants will receive a copy of the debriefing form, which provides further information about the study purpose, independent and dependent variables, local mental health resources, and contact information for the LPI. The debriefing form will be emailed to participants via McMaster Outlook using the email encryption function. If participants do not complete the study questionnaires, the debriefing form will be sent to participants after their study time slot has closed.

The data will be collected and stored through the secure online data collection platform REDCap, which is managed by St. Joseph's Healthcare Hamilton. REDCap is a secure, encrypted data collection platform that requires two-factor authentication for access to study data. REDCap is located within the secure internal SJHH network, and is protected by firewall software (Checkpoint software).

ELIGIBILITY:
Inclusion Criteria:

* 17 years of age or older
* Female
* Normal hearing with or without listening device

Exclusion Criteria:

* Currently diagnosed with an eating disorder
* Has received treatment for an eating disorder at any point in time

Min Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-09 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in measure of the Belief in Controlling Weight scale from baseline to post-intervention | Baseline (questionnaires administered prior to watching videos) and Post-Intervention (questionnaires administered after watching the videos) approximately 1 hour after completing baseline questionnaires.
  Weight Control Beliefs Questionnaire - Belief in Control over Weight (BCWeight) scale. This is a validated self-report measure of the individual's belief in personal control over weight.
  The minimum score is 9 (low belief in controlling weight) and the maximum score is 36 (high belief in controlling weight). A higher score has been associated with negative/worse outcomes.
Change in measure of the Belief in Controlling Lifestyle scale from baseline to post-intervention | Baseline (questionnaires administered prior to watching videos) and Post-Intervention (questionnaires administered after watching the videos) approximately 1 hour after completing baseline questionnaires.
  Weight Control Beliefs Questionnaire - Belief in Control over Lifestyle (BCLifestyle) scale. This is a validated self-report measure of the individual's belief in striving for a healthy lifestyle with acceptance of the resulting weight.
  The minimum score is 8 (low belief in striving for a healthy lifestyle with acceptance of resulting weight) and the maximum score is 32 (high belief in striving for a healthy lifestyle with acceptance of resulting weight). A higher score has been associated with positive/better outcomes.

SECONDARY OUTCOMES:
Change in measure of Self-Esteem from baseline to post-intervention | Baseline (questionnaires administered prior to watching videos) and Post-Intervention (questionnaires administered after watching the videos) approximately 1 hour after completing baseline questionnaires.
  Rosenberg Self-Esteem Scale. This is a validated self-report measure of self-esteem.
  The minimum score is 10 and the maximum score is 40. A higher score indicates higher self-esteem (positive/better outcome).
Change in measure of Intentions to engage in dietary restraint from baseline to post-intervention | Baseline (questionnaires administered prior to watching videos) and Post-Intervention (questionnaires administered after watching the videos) approximately 1 hour after completing baseline questionnaires.
  The Eating Disorder Examination Questionnaire - Restraint Sub-scale, modified to assess intentions to engage in dietary restraint rather than dietary restraint over the past 28 days. Items are otherwise identical to original scale, which is a well-validated self-report measure.
  The minimum score is 0 and the maximum score is 25. A higher score indicates greater intentions to engage in dietary restraint (negative/worse outcome).
Change in measure of Body Appreciation from baseline to post-intervention | Baseline (questionnaires administered prior to watching videos) and Post-Intervention (questionnaires administered after watching the videos) approximately 1 hour after completing baseline questionnaires.
  Body Appreciation Scale - 2. This is a well-validated self-report measure of positive attitudes towards one's body.
  The minimum score is 10 and the maximum score is 50. A higher score indicates greater appreciation for one's body (positive/better outcome).
Change in measure of Fear of Self-Compassion for Weight and Shape from baseline to post-intervention | Baseline (questionnaires administered prior to watching videos) and Post-Intervention (questionnaires administered after watching the videos) approximately 1 hour after completing baseline questionnaires.
  Fear of Self-Compassion for Weight and Shape Scale. This scale is based on the Fear of Self-Compassion Scale (a well-validated self-report measure) with items modified to measure a fear of self-compassion for one's weight and shape. Items are otherwise identical to the original scale and recent findings suggests the modified scale has maintained its psychometric properties.
  The minimum score is 15 and the maximum score is 75. A higher score indicates more fear of self-compassion for ones weight and shape (a negative/worse outcome).
Change in measure of Self-Compassion for Weight & Shape from baseline to post-intervention | Baseline (questionnaires administered prior to watching videos) and Post-Intervention (questionnaires administered after watching the videos) approximately 1 hour after completing baseline questionnaires.
  Self-Compassion for Weight & Shape Scale. This scale is based on the Self-Compassion scale (a well-validated self-report measure), modified to measure self-compassion for weight and shape. Items are otherwise identical to the original scale and recent findings suggest the modified scale retains good psychometric properties.
  The minimum score is 12 and the maximum score is 60. A higher score indicates more self-compassion for ones weight and shape (a positive/better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Michele Laliberte, PhD, Principal Investigator — St. Joseph's Healthcare Hamilton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tylka TL, Wood-Barcalow NL. The Body Appreciation Scale-2: item refinement and psychometric evaluation. Body Image. 2015 Jan;12:53-67. doi: 10.1016/j.bodyim.2014.09.006. Epub 2014 Oct 21. PMID 25462882
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Craig C, Marshall A, Sjostrom M, Bauman A, Lee P, Macfarlane D, Lam T, & Stewart S. International physical activity questionnaire-short form. Journal of American College Health. 2017; 65(7): 492-501.
- [Background] Laliberte MM, Newton M, McCabe R, & Mills JS. Controlling Your Weight Versus Controlling Your Lifestyle: How Beliefs about Weight Control Affect Risk for Disordered Eating, 10534_2006_9060_Fig3_HTML.gif Dissatisfaction and Self-esteem. Cognitive Therapy and Research. 2007; 31(6): 853-869.
- [Background] Rosenberg M. Society and the Adolescent Self-Image (Revised edition). Wesleyan University Press. 1989.